



Mr. Alex Green

John Radcliffe Hospital

01865 741166

Study Code: Site ID Code: Participant identification number:

## **CONSENT FORM**

## <Study Title>: Cerebral Signature for pain perception and modulation

Name of Researcher: Dr Tariq Parker, MBBS, Msc If you agree, please initial box

| 1. | I confirm that I have read the information sheet dated 28/05/2018 (version 7) for this study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. |
|---|---|
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. |
| 3. | I understand that relevant sections of my medical notes (if relevant) and data collected during the study may be looked at by individuals from University of Oxford, from regulatory authorities and from the NHS Trusts, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. |
| 4. | I understand that the information collected about me may be used in an anonymous form to support other research in the future. It will not be possible for me to be identified by it. |
| 5. | I understand that this is a research scan that is not useful for medical diagnosis, and that scans are not routinely looked at by a doctor. If a concern is raised about a possible abnormality on my scan, I will only be informed if a doctor thinks it is medically important such that the finding has clear implications for my current or future health. |
| 6. | I agree to take part in this study. |

Pain Study Consent form Version/Date: Version 7/ 28/05/2018
The Cerebral Signature for Pain Perception and Its modulation
Mr. Alex Green REC Reference number: 13/SC/0298

| 7. I agree to be contacted about ethically approved research studies for which I may be suitable. I understand that agreeing to be contacted does not oblige me to participate in any further studies. | | |
|---|---|---|
| me to participate in any fu | The to participate in any further studies. | |
| Name of Participant | Date | Signature |
| Name of Person taking<br>Consent | Date | Signature |

<sup>\*1</sup> copy for participant; 1 copy for researcher site file; 1 (original) to be kept in medical notes (if participant is a patient).